CLINICAL TRIAL: NCT03973775
Title: A Double Blind, Two Arm, Multicenter, Randomized, Parallel Group, Bioequivalence Study With Clinical Endpoints to Evaluate the Safety and Therapeutic Equivalence of Permethrin Cream 5% & Elimite™ in Subjects With Scabies
Brief Title: A Bioequivalence Study With Clinical Endpoints to Evaluate the Safety and Therapeutic Equivalence of Permethrin Cream 5% & Elimite™ in Subjects With Scabies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Saptalis Pharmaceuticals LLC (Industry)
Collaborators: bioRASI, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SP-2992
Record Dates: First submitted 2019-05-30; First posted 2019-06-04 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Scabies
MeSH Terms: conditions — Scabies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The Study Team consisted of blinded and unblinded teams. The blinded team consists of the Principal investigator(s) and their designee(s). This team includes trained study personnel who are experienced at finding scabies mites in skin lesions. Blinded team members completed informed consent/assent, screen for inclusion/exclusion criteria, enroll subjects, collect demographic information, perform the pre- and post-treatment evaluations and complete the Case Report Forms (CRFs). The unblinded team members consists of the dedicated study pharmacist and/or their designee(s).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Drug Treatment Arm (Experimental): Permethrin Cream 5%, Saptalis Pharmaceuticals, LLC
  Interventions: Drug: Permethrin Cream 5%
- Reference Drug Treatment Arm (Active Comparator): Elimite™ (Permethrin Cream 5%), Prestium Pharma, Inc.
  Interventions: Drug: Permethrin Cream 5%

INTERVENTIONS:
Drug: Permethrin Cream 5% — Patients will be assigned to the test product Permethrin Cream 5% to the Reference Listed Drug Product Elimite cream.

SUMMARY:
This phase III study was conducted to establish the clinical bioequivalence of Permethrin Cream 5% and Elimite™ in the treatment of scabies following a single application.

DETAILED DESCRIPTION:
A Double Blind, Two Arm, Multicenter, Randomized, Parallel Group Bioequivalence Study with Clinical Endpoints to Evaluate the Safety and Therapeutic Equivalence of, Permethrin Cream 5% (Manufactured by Saptalis Pharmaceuticals, LLC) & Elimite™ (Permethrin Cream 5%, manufactured for Prestium Pharma, Inc.) in Subjects with Scabies.

The objectives of this study are:

Primary Objective: To establish the clinical bioequivalence of Permethrin Cream 5% (manufactured by Saptalis Pharmaceuticals, LLC) and Elimite™ (Permethrin Cream 5%, manufactured for Prestium Pharma, Inc.) in the treatment of scabies (Sarcoptes scabiei) following a single application.

Secondary Objective: To compare the safety and tolerability between the study drugs.

ELIGIBILITY:
Inclusion Criteria:

* Subjects and/or parent/guardian must have understood and signed appropriately administered informed consent/assent in their own language
* Healthy male and non-pregnant/non-lactating female subjects aged 2 months to 65 years diagnosed with scabies
* Must have dermatological evidence of active scabies (burrows, erythematous papules, etc.) confirmed by recovery of live Sarcoptes scabiei (the Principal investigator or trained and experienced Study Team examines the specimen(s) under magnification to verify the identity and viability of the scabies mite, ova, or mite feces at the site)
* The youngest subject (with scabies infestation as defined above) from each household is considered the index or primary subject of the household for evaluation of the primary endpoint. Other members of the household and close contacts are enrolled in the study as Secondary subjects and evaluated for all safety parameters (not included in primary endpoint analysis). Secondary subjects that are confirmed to have dermatological evidence of scabies should receive the same study treatment as the Index subject
* Must be available and willing to report for follow up visits
* Is otherwise healthy, well-nourished, non-febrile and not suffering from an infection likely to require systemic antibiotic or topical therapy. These criteria will be ascertained during screening by the Principal investigator
* Must agree not to use other scabicides or other medications likely to affect the evaluation of their response to scabies treatment
* If female of childbearing potential, willing to use an acceptable method of birth control, should be stable for 3 months prior to screening and throughout the study
* Must be willing to follow the procedures to decrease infestation: Clothes and bed linens that were in contact with the subjects, their household members and close contacts during the previous 48 to 72 hours will be machine washed at 60°C and machine dried the day after the first treatment. For materials that cannot be laundered, insecticide powder or aerosolized insecticide may be used, or the items may be kept in a sealed bag for at least 48 to 72 hours.

Exclusion Criteria:

* Subject or parent/guardian has not signed informed consent/assent
* Pregnant females, lactating females or females planning for a pregnancy
* Females of childbearing potential who do not agree to utilize an adequate method of contraception
* Known history of irritation or sensitivity to parasiticides
* Skin conditions that could make it difficult to evaluate the extent of an infestation or would present a problem in the evaluation of response to therapy (e.g. atopic dermatitis, eczema, contact dermatitis, lichen planus, papular urticaria, seborrheic dermatitis).
* Use within 4 weeks of baseline visit (1) immunomodulators (2) systemic medications that suppress the immune system (3) topical or oral parasiticides.
* Use within 2 weeks of baseline visit (1) topical steroids (2) topical or systemic antibiotics
* Has crusted scabies • Known allergy or hypersensitivity to permethrin, any synthetic pyrethroid or pyrethrin, plants in the Asteraceae/Compositae family (e.g. chrysanthemums, ragweed, marigolds, and daisies)
* Subjects whose household members and close contacts refuse treatment.
* Subjects with greater than 5 infested household members and close contacts
* Subjects whose sexual contacts do not agree to restrict prolonged skin to skin contact with non-household members during the study period
* Subjects with a household member less than 2 months of age
* Suffers from a renal or hepatic impairment
* Has been treated for scabies by any form of scabies treatment whether prescription, over-the-counter or a home remedy within a month prior to their screening visit
* Had received or used an investigational new drug within the month immediately preceding the screening
* Is receiving any medication likely to mask or modify scabies
* Will not be available for follow up visits
* Has other cutaneous conditions which might be confused with scabies
* Seriously immune suppressed subjects
* Has been previously empaneled in this study

Ages: 2 Months to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2018-12-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the proportion of index subjects in the Per Protocol (PP) population in each treatment group with treatment cure when examined at Visit 4 (Day 28 ± 2 Days). | Day 28 ± 2 Days
  Cure is defined as demonstration of clinical cure (all clinical findings have completely resolved, including inflammatory/non-inflammatory lesions) and microscopic cure (demonstration of the absence of mites, ova, and/or mite feces) on Day 28. Negative microscopy can be declared if no mites, ova, or mite feces is found from a minimum of 3 skin scrapings from previously affected sites.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Universal Biopharma Research Institute Inc., Dinuba, California
  - Long Beach Clinical Trials Services, Inc., Long Beach, California
  - Havana Research Institute, Pasadena, California
  - SouthCoast Research Center, Inc (Clinical Site & Drug Shipment Facility), Miami, Florida
  - West Houston Clinical Research Service, Houston, Texas

REFERENCES:
- [Background] Goldust M, Babae Nejad S, Rezaee E, Raghifar R. Comparative trial of permethrin 5% versus lindane 1% for the treatment of scabies. J Dermatolog Treat. 2013 Jan 20. doi: 10.3109/09546634.2012.723122. Online ahead of print. PMID 22905702
- [Background] Oliva ME, Rekha A, Yellin A, Pasternak J, Campos M, Rose GM, Babinchak T, Ellis-Grosse EJ, Loh E; 301 Study Group. A multicenter trial of the efficacy and safety of tigecycline versus imipenem/cilastatin in patients with complicated intra-abdominal infections [Study ID Numbers: 3074A1-301-WW; ClinicalTrials.gov Identifier: NCT00081744]. BMC Infect Dis. 2005 Oct 19;5:88. doi: 10.1186/1471-2334-5-88. PMID 16236177
- See also: Mechanism of action — http://www.drugbank.ca/drugs/db04930
- See also: Related Info — https://pubchem.ncbi.nlm.nih.gov/compound/Permethrin
- See also: Related Info — https://dailymed.nlm.nih.gov/dailymed/fda/fdaDrugXsl.cfm?setid=aa294be5-90154f6a-8a92-a71a2b22d1b2&type=display